CLINICAL TRIAL: NCT03324802
Title: A Phase III Trial of Hypofractionated Radiotherapy to the Whole Breast Alone After Breast Conserving Surgery
Brief Title: Hypofractionated Radiation Therapy in Preventing Recurrence in Patients With Breast Cancer After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MC1635; NCI-2017-01944 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1635 (Other: Mayo Clinic in Arizona); NCT03339934 (obsolete NCT alias)
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 2 (hypofractionated radiation therapy, 5 fractions) (Experimental): Within 12 weeks of breast cancer surgery or adjuvant chemotherapy, patients undergo hypofractionated radiation therapy in 5 daily fractions for 5 days.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment
- Arm I (radiation therapy, 15 fractions) (Experimental): Within 12 weeks of breast cancer surgery or adjuvant chemotherapy, patients undergo standard radiation therapy in 15 daily fractions for 10 days.
  Interventions: Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
  Arms: Arm 2 (hypofractionated radiation therapy, 5 fractions)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — hypofractionated radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm I (radiation therapy, 15 fractions)

SUMMARY:
This randomized phase III trial studies how well hypofractionated radiation therapy works in preventing the return of tumor cells in breast cancer patients following surgery. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 24-month complication rate of 5 fraction whole radiotherapy +/- concurrent boost as compared to 15 fraction radiotherapy +/- sequential boost.

SECONDARY OBJECTIVES:

I. To evaluate acute and late toxicity. II. To estimate the 5-year locoregional control, invasive disease-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To evaluate fatigue, and other patient-reported outcomes. II. To evaluate clinical features, treatment technique, dose-volume parameters, histologic and genetic variants associated with fair and poor cosmetic outcomes or unplanned surgical intervention.

III. To evaluate the costs and comparative effectiveness of treatment. IV. Compare the use of photon therapy with spot scanning proton therapy in two different hypo-fractionated whole breast schemas.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Within 12 weeks of breast cancer surgery or adjuvant chemotherapy, patients undergo radiation therapy in 15 daily fractions for 10 days.

ARM II: Within 12 weeks of breast cancer surgery or adjuvant chemotherapy, patients undergo hypofractionated radiation therapy in 5 daily fractions for 5 days.

After completion of study treatment, patients are followed up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast cancer
* Pathologic stage T0-T3N0-N1M0
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Able to and provides Institutional Review Board (IRB) approved study specific written informed consent
* Study entry must be within 12 weeks of last surgery (breast or axilla) or last chemotherapy (if applicable)
* Able to complete all mandatory tests
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Fair, good or excellent cosmesis, as determined by trained nurse assessment using the Harvard Cosmetic Scale
* Radiotherapy must begin within 12 weeks of the last breast cancer surgery or the last dose of adjuvant chemotherapy
* Breast conserving surgery and indications for whole breast radiotherapy

Exclusion Criteria:

* Medical contraindication to receipt of radiotherapy
* Severe active co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or providing informed consent
* Active systemic lupus or scleroderma
* Pregnancy
* Prior receipt of ipsilateral breast or chest wall radiation
* Positive margins on ink after definitive surgery either for ductal carcinoma in situ (DCIS) or invasive cancer
* History of non-breast malignancies (except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin) within 5 years prior study entry
* Recurrent breast cancer
* Indications for comprehensive regional nodal irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Vargas, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Radiation Therapy, 15 Fractions): Within 12 weeks of breast cancer surgery or adjuvant chemotherapy, patients undergo standard radiation therapy in 15 daily fractions for 10 days.
  Quality-of-Life Assessment: Ancillary studies
  Radiation Therapy: hypofractionated radiation therapy
- Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions): Within 12 weeks of breast cancer surgery or adjuvant chemotherapy, patients undergo hypofractionated radiation therapy in 15 daily fractions for 10 days.
  Quality-of-Life Assessment: Ancillary studies
  Hypofractionated Radiation Therapy: Undergo hypofractionated radiation therapy
Period: Overall Study
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Started | 54 | 53
Completed | 54 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions) | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (7.7) | 62.9 (9.3) | 62.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 50 | 49 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 54 | 53 | 107
Study breast [Count of Participants; unit: Participants]
  Left | 28 | 30 | 58
  Right | 26 | 23 | 49
Bilateral disease [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 54 | 52 | 106
Multiple lesions [Count of Participants; unit: Participants]
  Yes | 5 | 12 | 17
  No | 49 | 41 | 90

OUTCOME MEASURES:

1. Primary Outcome: Complication Rate, Defined as the Percentage of Women Who Develop Grade 3 or Higher Late Adverse Event and/or Deterioration of Cosmesis From Excellent/Good to Fair/Poor or From Fair to Poor
Description: The complication rate will be reported by arm.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
Participants | 2 | 3

2. Secondary Outcome: Cause-specific Survival
Description: Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Estimates will be given for one year with 95% CIs. Comparison between arms will employ a log-rank test.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
percentage of patients | 100 [NA to NA] — 95% CI not able to be calculated since all patients were alive at 1 year | 100 [NA to NA] — 95% CI not able to be calculated since all patients were alive at 1 year
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 1.0, Log Rank

3. Secondary Outcome: Overall Survival
Description: Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Estimates will be given for one year along with 95% CIs. Comparison between arms will employ a log-rank test.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
percentage of patients | 100 [NA to NA] — 95% CI not able to be calculated since all patients were alive at 1 year | 100 [NA to NA] — 95% CI not able to be calculated since all patients were alive at 1 year
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 1.0, Log Rank

4. Secondary Outcome: Number of Patients Experiencing Distant Recurrence
Description: Distant recurrence defined as metastatic cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
Participants | 0 | 0

5. Secondary Outcome: Number of Patients Experiencing Acute (Grade 3+) Adverse Events (AEs)
Description: The maximum grade for each type of acute (grade 3+) AE will be recorded for each patient. Data will be summarized as frequencies and relative frequencies by treatment arm. The relationship of the adverse event(s) to the study treatment will be taken into consideration. Number of patients experiencing one or more grade 3+ events will be compared between arms using chi-squared tests. Adverse events were assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
Participants | 1 | 0
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 0.320, Chi-squared

6. Secondary Outcome: Number of Patients Experiencing Grade 3+ Late Adverse Events
Description: The maximum grade for each type of late AE will be recorded for each patient. Data will be summarized as frequencies and relative frequencies by treatment arm. The relationship of the adverse event(s) to the study treatment will be taken into consideration. Number of patients experiencing one or more grade 3+ late AEs will be compared between arms using chi-squared tests.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
Participants | 1 | 4
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 0.163, Chi-squared

7. Secondary Outcome: Invasive Disease-free
Description: Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Median invasive disease-free time will be given along with standard error. Comparison between arms will employ a log-rank test.
Time Frame: 5 years
Measure: Median (Standard Error); unit: years
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
years | 2.9569 (0.0225) | 3.4743 (0.0298)
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 0.97, Log Rank

8. Secondary Outcome: Percent of Patients With Locoregional Recurrence
Description: The cumulative incidence of locoregional recurrence will be estimated using a competing risks method by treatment arm. The competing risks will be distant breast cancer recurrence and death. Comparison between arms will employ Fine-Gray regression. Locoregional recurrence is clinically diagnosed invasive breast cancer in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast at 5 years.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
percentage of patients | 2.3 [0.17 to 10] | 5.8 [1.0 to 17]
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 0.5, Gray Test P-value

9. Secondary Outcome: Disease-Free Survival
Description: Will be estimated with a Kaplan-Meier estimator and curve by treatment arm. Median disease free survival time and standard error will be estimated. Comparison between arms will employ a log-rank test.
Time Frame: 5 years
Measure: Median (Standard Error); unit: years
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
Number analyzed (Participants) | 54 | 53
years | 2.9569 (0.0225) | 3.17 (0.0282)
Statistical Analysis 1: Comparison: Arm 1 (Radiation Therapy, 15 Fractions) vs Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions); Test type: Superiority; p = 0.54, Log Rank

10. Other Pre Specified Outcome: Patient Reported Outcomes/Quality of Life
Description: The subscales of the Breast Cancer Treatment Outcomes Scale (BCTOS), elements from Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), and other patient reported measures such as fatigue, breast pain, breast shape, and arm related morbidity outlined in the appendix will be summarized as the mean +/- standard deviation and median (minimum value, maximum value). Mixed models will be used to estimate changes at fixed time points.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Patient Reported Outcomes/Quality of Life
Description: The subscales of the Breast Cancer Treatment Outcomes Scale (BCTOS), elements from Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE), and other patient reported measures such as fatigue, breast pain, breast shape, and arm related morbidity outlined in the appendix will be summarized as the mean +/- standard deviation and median (minimum value, maximum value). Mixed models will be used to compare outcomes between arms.
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patient Self-reported Cosmesis
Description: Will evaluate fatigue, breast pain, arm function. The values of the cosmesis instruments (patient self-reported and panel-assessed) will be summarized with the frequencies and confidence intervals of fair or poor cosmesis events at baseline, 2 years, and 5 years by treatment arm. Comparisons between arms will employ chi-squared tests.
Time Frame: Baseline up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Arm 1 (Radiation Therapy, 15 Fractions) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions)
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 50/54 | 51/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Radiation Therapy, 15 Fractions) (N=54) | Arm 2 (Hypofractionated Radiation Therapy, 5 Fractions) (N=53)
Dermatitis radiation (Injury, poisoning and procedural complications) | 43 (48) | 36 (44)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (6) | 5 (7)
Lymphedema (Vascular disorders) | 19 (42) | 20 (48)
Pain (General disorders) | 26 (56) | 23 (51)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 29 (48) | 29 (55)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 4 (8) | 9 (13)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 12 (20) | 12 (19)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/02/NCT03324802/Prot_SAP_000.pdf